CLINICAL TRIAL: NCT06344975
Title: A Phase 1/2, Randomized, Placebo-Controlled, Double-Blind, Dose-Finding, First-in-Human Study of Respiratory Syncytial Virus (RSV) mRNA Vaccine STR-V003 in Healthy Adults
Brief Title: A Study to Describe the Safety and Immunogenicity of a Respiratory Syncytial Virus Vaccine STR-V003 in Healthy Adults
Acronym: STR-V003
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Starna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: Starna Therapeutics
Record Dates: First submitted 2024-03-25; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort1 (Experimental): Cohort 1: Dose A in Younger/older Adults
  Single injection of Dose A of STR-V003 or placebo on Day 0.
  Interventions: Biological: STR-V003/Placebo
- Cohort2 (Experimental): Cohort 2: Dose B in Younger/older Adults
  Single injection of Dose B of STR-V003 or placebo on Day 0.
  Interventions: Biological: STR-V003/Placebo
- Cohort3 (Experimental): Cohort 3: Dose C in Younger/older Adults
  Single injection of Dose C of STR-V003 or placebo on Day 0.
  Interventions: Biological: STR-V003/Placebo
- Cohort4 (Experimental): Cohort 4: Dose B in Younger/older Adults
  Two injections of Dose B of STR-V003 or placebo on Day 0 and Day21.
  Interventions: Biological: STR-V003/Placebo

INTERVENTIONS:
Biological: STR-V003/Placebo — IM

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose escalation and two-dose study in healthy adults. This study will be conducted in healthy men and women ≥18 years old to assess the safety, tolerability and immunogenicity of STR-V003. This trial consists of two parts: Part A and Part B.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and willing to sign the ICF.
2. Healthy male and female subjects, non-smokers defined as having abstained from tobaccoornicotine containing products (e.g., cigarettes, chewing tobacco, snuff, nicotine patches,and electronic cigarettes) in the 6 months prior to the Screening.
3. Must be ≥18 years of age.
4. With no significant medical history, and in good health as determined by detailed medical history (neurological, endocrinal, cardiovascular, pulmonary, hematological, immunologic,psychiatric, gastrointestinal, renal, hepatic, and metabolic disease), full physicalexamination, vital signs, 12-lead electrocardiogram (ECG), urinalysis and laboratory tests at screening.

   4.1) Abnormal laboratory or vital signs results may be repeated once if abnormal result is observed at the initial reading.

   4.2) Abnormalities found in the ECG may need to be confirmed by repeated measurements.
5. Subjects must have adequate organ function according to the following laboratory values:

   5.1) Bone marrow function (absolute neutrophil count ≥ 1500/mm3 and platelet count ≥100,000/mm3) 5.2) Adequate liver function [alanine aminotransferase (ALT) ≤ 1.5 × upper limit normal(ULN) and alkaline phosphatase ≤ 1.5 × ULN, total bilirubin ≤ 1.5 mg/dL] 5.3) Adequate renal function creatinine clearance 60 mL/min based on Cockcroft-Gaultequation, or serum creatinine level ≤ 1.5 times the ULN
6. Be a female of non-childbearing potential [i.e., physiologically incapable of becoming pregnant, including any female who is 2 years post-menopausal and have an FSH > 40mIU/mL, or surgically sterile (defined as having a bilateral oophorectomy, hysterectomy or tubal ligation)] or agree to one of the following to prevent pregnancy.
7. If a woman of childbearing potential, she must have a negative serum pregnancy test at screening:

   7.1) Practicing abstinence. 7.2) If a sexually active woman of childbearing potential (sexually active with a non-sterile male partner) she must agrees to prevent pregnancy by using double methods of contraception as until at least 6 months after the last dose of the investigational product.
8. Male subjects who are not vasectomized for at least 6 months and who are sexually active with a non-sterile female partner must agree to use double methods of contraception as and must not donate sperm until 6 months after the last dose during their study participation period:
9. Body mass index (BMI) 18.0-30.0 kg/m2 documented at screening and day-1.
10. Blood pressure ≤ 139/89 mm Hg.
11. Subjects are able to follow the study protocol and complete the trial.

Exclusion Criteria:

1. Pregnancy or lactation.
2. History or presence of conditions which, in the judgment of the Investigator, are known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
3. History of any clinically significant medical illness or medical disorders the Investigator considers should exclude the subject, including (but not limited to) immune deficient state; neuromuscular, hematological, cardiac, vascular, metabolic, endocrine, rheumatologic,respiratory, hepatic, gastrointestinal, neurological, neoplastic, dermatological, renal, urinary tract, or psychiatric disease, hypertension, osteoarthritis or ophthalmological disorders.
4. Clinically significant abnormalities on ECG, including a QT corrected according to Fridericia's formula (QTcF) interval > 450 msec (males) or > 470 msec (for females).
5. History of surgery or major trauma within 6 months prior to study screening.
6. History of any significant hypersensitivity reaction to medications, including manifestations suggestive of anaphylaxis.
7. History or presence of any active infection within 14 days, or an infection requiring prescription therapy or hospitalization within 30 days of enrollment.
8. History of alcohol abuse, illicit drug use, physical dependence on any opioid, or any history of drug abuse or addiction within 12 months of Screening.
9. Use of prescription medications within 30 days or 5 half-lives, whichever is longer, prior to administration of the study drug.

   9.1) Hormonal birth control will be permitted.
10. Use of OTC drugs (including herbal preparations) within 14 days or 5 half-lives (if known),whichever is longer, prior to administration of the study drug.
11. Received a vaccination within 30 days prior to administration of the study drug.
12. Any investigational drugs or participated in any clinical study within 30 days or 5 half-lives(if known), whichever is longer, prior to administration of the study drug in this study.
13. Significant blood loss (> 450 mL) or has donated 1 or more units of blood or plasma within 6 weeks prior to study participation.
14. Strenuous activity (as assessed by the Investigator) within 48 hours prior to CRU admission.
15. Consumption of alcohol, xanthine (i.e., chocolate), caffeine-containing food or beverages within 3 days prior to CRU admission. Consumption of alcohol is restricted to within 48hours of follow-up visits.
16. Positive test for HIV-1 or HIV-2 antibodies, or positive test for HBV or HCV consistent with current infection. Confirmatory tests will be allowed at the discretion of the Investigator to rule out false positives.
17. History or presence of any bleeding disorders, or symptoms suggestive of a bleeding disorder.
18. Unwilling or unlikely to comply with the requirements of the study.
19. Immunocompromised individuals and those with a history of autoimmune disease.
20. Increased risk for severe RSV infection
21. Positive serological test for SARS-CoV-2 IgM and/or IgG at the screening visit, and a SARS-CoV-2 nucleic acid amplification test-positive nasal swab within 24 h before study vaccination.
22. History of severe adverse reaction associated with a vaccine and/or severe allergic reaction(e.g., anaphylaxis) to any component of the investigational product(s), including natural rubber latex.
23. Previous clinical or microbiological diagnosis of RSV, receipt of medications intended to prevent RSV, previous vaccinations including any investigational or licensed RSV vaccine or other related RSV product.
24. Any participant who is acutely ill or febrile (body temperature ≥ 38.0°C/100.4°F) within 48hours prior to or on the date of vaccination. The participant should not be included in the study until the condition has resolved for at least 2 consecutive days before the vaccination day.
25. Any participant who has received or plans to receive an mRNA vaccine within 60 days of study vaccination.
26. Any participant with a history of myocarditis or pericarditis.
27. Any participant with history of an immune-mediated neurological disease, including Guillain-Barré Syndrome (GBS).
28. Have a screening abnormality that is > Grade 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Immediate unsolicited AEs for 30 minutes post-vaccination | 30 minutes
  Percentage of Participants With Immediate unsolicited AEs Through 30 minutes After Initial Vaccination
Solicited injection site (local) and systemic reactions for 7 days postvaccination. | 7 days
  Percentage of Participants With Solicited injection site (local) and systemic reactions for 7 days After Initial Vaccination
Unsolicited AEs for 28 days postvaccination | 28 days
  Percentage of Participants With Unsolicited AEs for 28 days After Initial Vaccination
Medically attended adverse events (MAAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) for the entire study duration | 12 months
  Percentage of Participants With Medically attended adverse events (MAAEs), serious adverse events (SAEs), and adverse events of special interest (AESIs) for the entire study duration

IPD SHARING:
Plan to Share IPD: No